CLINICAL TRIAL: NCT02174978
Title: Phase 1 Clinical Trial With Controlled Human Malaria Infection (CHMI) Open-label Dose Safety, Reactogenicity, Immunogenicity, and Efficacy of the Vaccine Candidate Plasmodium Falciparum Malaria Protein (FMP012), Administered Intramuscularly With AS01B Adjuvant System in Healthy Malaria-Naïve Adults
Brief Title: Phase 1 Clinical Trial With Controlled Human Malaria Infection (CHMI) to Evaluate the Safety and Efficacy of the Plasmodium Falciparum Vaccine Candidate FMP012 Administered Intramuscularly With AS01B Adjuvant System in Healthy Malaria-Naïve Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); United States Agency for International Development (USAID) (U.S. Federal Agency); Military Infectious Diseases Research Program (MIDRP) (Network); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S-14-02
Record Dates: First submitted 2014-06-11; First posted 2014-06-26 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Malaria
Keywords: Malaria vaccine
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1: 10 µg FMP012 adjuvanted AS01B (Experimental): FMP012 with AS01B adjuvant system: 10 µg FMP012 antigen reconstituted with 500 µL AS01B adjuvant to equal 0.5 mL final volume. Doses administered intramuscular at week 0, 4, 8, and 24. On week week 27, there is a P falciparum Controlled Human Malaria Infection (CHMI) challenge.
  Interventions: Biological: FMP012 with AS01B adjuvant system; Other: P falciparum Controlled Human Malaria Infection (CHMI)
- Group 2: 30 µg FMP012 adjuvanted AS01B (Experimental): FMP012 with AS01B adjuvant system: 30 µg FMP012 antigen reconstituted with 500 µL AS01B adjuvant to equal 0.5 mL final volume administered intramuscular at week 2, 6, 10, and 24. On week week 27, there is a challenge with P falciparum Controlled Human Malaria Infection (CHMI).
  Interventions: Biological: FMP012 with AS01B adjuvant system; Other: P falciparum Controlled Human Malaria Infection (CHMI)
- Infectivity control (Other): Non-immunized infectivity control challenged with P falciparum Controlled Human Malaria Infection (CHMI)
  Interventions: Other: P falciparum Controlled Human Malaria Infection (CHMI)

INTERVENTIONS:
Biological: FMP012 with AS01B adjuvant system — Candidate malaria vaccine based on the recombinant protein FMP012, which is Escherichia coli-expressed Plasmodium falciparum cell-traversal protein for ookinetes and sporozoites (PfCelTOS)
  Other Names: FMP012 antigen adjuvanted with AS01B
  Arms: Group 1: 10 µg FMP012 adjuvanted AS01B; Group 2: 30 µg FMP012 adjuvanted AS01B
Other: P falciparum Controlled Human Malaria Infection (CHMI)

SUMMARY:
The proposed study is a Phase 1 study with controlled human malaria infection (CHMI) designed primarily to evaluate the safety of the FMP012 combined with AS01B adjuvant system. AS01B is a proprietary current good manufacturing practices (cGMP) grade adjuvant manufactured by GlaxoSmithKline (GSK) Biologicals. It is a formulation based on liposomes mixed with the immunostimulants monophosphoryl lipid (MPL) and Quillaja saponaria (QS)-21. The immunogenicity and efficacy of this new candidate vaccine will be evaluated in addition to safety.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (male or non-pregnant, non-lactating female) 18 to 50 years of age (inclusive) at the time of screening
* If the subject is female,

  * Non-childbearing potential (ie, either surgically sterilized or one year post-menopausal), abstinent or using adequate contraceptive precautions (eg, intrauterine contraceptive device; oral contraceptives; diaphragm or condom in combination with contraceptive jelly, cream or foam; Norplant® or Depo-Provera®) during this study and must agree to continue such precautions until three months after challenge
  * A negative pregnancy test at the time of enrollment
* Free of significant health problems as established by medical history, laboratory, and clinical examination before entering the study
* Subjects must have low cardiac risk factors according to the National Health and Nutrition Examination Survey (NHANES) I criteria, medical history and family history, blood pressure measurements, and a normal or normal variant ECG
* Available to participate and reachable by phone for duration of study (approximately 8-14 months) and reachable by phone at the 6 month post Controlled Human Malaria Infection (CMHI) follow-up
* No plans to travel to outside the Washington DC area between the day of challenge and either completion of treatment course (post-challenge) or, if subject remains uninfected, 28 days post-challenge
* No plans to travel to a malaria endemic area during the course of the study
* Written informed consent must be obtained from the subject before screening procedures are performed
* Subjects must score at least 80% correct on a multiple-choice quiz that assesses their understanding of this study
* If a subject is active duty military, he or she must obtain approval from his or her supervisor per Walter Reed Army Institute of Rese (WRAIR) Policy 11-45

Exclusion Criteria:

* Any history of malaria infection
* History of travel to P falciparum endemic areas in the 3 months prior to day of first vaccination (Vaccination Groups) or day of challenge (Infectivity Control Group)
* Any history of receiving a malaria vaccine
* Receipt of any licensed vaccine within 7 days prior to first vaccination (Note: subjects are encouraged to get recommended licensed preventive vaccinations during the course of the study but are requested to schedule any routine preventive vaccinations for at least 7 days before or after a scheduled FMP012/AS01B vaccination day)
* History of receipt of malaria prophylaxis during the 2 months prior to day of first vaccination (Vaccination Groups) or day of challenge (Infectivity Control Group)
* History of use of any antibiotics with significant antimalarial activity (examples include tetracycline, doxycycline, clindamycin, azithromycin, and sulfa drugs) during the course of the study period (period starting one month prior to challenge, Infectivity Control Group)
* Use of any investigational or non-registered drug or vaccine within 30 days preceding the first dose of study vaccine or planned use during the study period.
* Any history of allergic reaction or anaphylaxis to previous vaccination (Vaccination Groups)
* Allergy to egg protein (Vaccination Groups)
* Pregnant (positive β-human chorionic gonadotropin test, β-HCG) or lactating female at screening or plans to become pregnant or breastfeed from the time of enrollment until three months after challenge
* Allergy to antimalarial drugs or use of medications known to interact with chloroquine (CQ)
* Significant (eg, systemic) hypersensitivity reactions to mosquito bites (local hypersensitivity reactions at the site of mosquito bites are not an exclusion criterion)
* History of sickle cell disease
* History of psoriasis or porphyria
* History of splenectomy
* Any confirmed or suspected immunodeficiency, including HIV infection
* Administration of chronic (defined as more than 14 days) immunosuppressive drugs or other immune-modifying drugs within 6 months of vaccination
* History of autoimmune disease
* Family history of congenital or hereditary immunodeficiency
* Acute or chronic, clinically significant, pulmonary, cardiovascular, endocrine, hepatic, or renal functional abnormality, as determined by history, physical examination, or laboratory evaluation
* Chronic or active neurologic disease including seizure disorder and chronic migraine headaches
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or any planned administration during the study period
* Any abnormal baseline laboratory screening tests to include:

  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) above normal range,
  * Creatinine above normal range,
  * Hemoglobin out of normal range,
  * Platelet count out of normal range, or
  * Total white blood cell (WBC) count out of normal range
* Seropositive for HIV or Hepatitis C virus (HCV) or hepatitis B surface antigen (HBsAg) positive
* Hepatomegaly, right upper quadrant abdominal pain or tenderness
* An abnormal baseline screening ECG suggestive of cardiac disease as determined by a clinical investigator
* Suspected or known current alcohol or drug abuse as determined from the medical history or by physical examination
* Any other significant finding that in the opinion of the PI would increase the risk of having an adverse outcome from participating in this study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Number of solicited adverse events (AE) | 7 days after each vaccination
Number of unsolicited AEs | 28 days after each vaccination
Occurrence of serious adverse events (SAE) at any time during the study period (enrollment to final follow-up visit) | 12 months after vaccination

SECONDARY OUTCOMES:
Anti-FMP012 antibody titers in serum | 12 months
Time to parasitemia by blood smear after the P falciparum challenge | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jason W Bennett, LTC, MC, Principal Investigator — Malaria Vaccine Branch, Military Malaria Research Program, WRAIR
Locations (1):
- Clinical Trials Center, WRAIR, Silver Spring, Maryland, United States